CLINICAL TRIAL: NCT03123185
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 705564 (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design) and Food Effect on a Tablet Formulation of BI 705564 (Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Design) in Healthy Male Subjects
Brief Title: Safety and Pharmacokinetics of Single Rising Doses of BI 705564 and Food Effect on BI 705564 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1408-0001; 2017-000324-98 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Placebo matching BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: Placebo
- Placebo matching BI 705564 fed (SRD part) (Experimental)
  Interventions: Drug: Placebo
- 1 milligram (mg) BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 3 mg BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 10 mg BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 20 mg BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 40 mg BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 80 mg BI 705564 fasted (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Reference)
- 20 mg BI 705564 fed (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Test)
- 40 mg BI 705564 fed (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Test)
- 80 mg BI 705564 fed (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Test)
- 160 mg BI 705564 fed (SRD part) (Experimental)
  Interventions: Drug: BI 705564 (Test)
- BI 705564 10 mg fasted/ BI 705564 10 mg fed (FE Part) (Experimental)
  Interventions: Drug: BI 705564 (Test); Drug: BI 705564 (Reference)
- BI 705564 10 mg fed/ BI 705564 10 mg fasted (FE Part) (Experimental)
  Interventions: Drug: BI 705564 (Test); Drug: BI 705564 (Reference)

INTERVENTIONS:
Drug: Placebo — Tablet and solution formulation
  Arms: Placebo matching BI 705564 fasted (SRD part); Placebo matching BI 705564 fed (SRD part)
Drug: BI 705564 (Test) — Fed state
  Arms: 160 mg BI 705564 fed (SRD part); 20 mg BI 705564 fed (SRD part); 40 mg BI 705564 fed (SRD part); 80 mg BI 705564 fed (SRD part); BI 705564 10 mg fasted/ BI 705564 10 mg fed (FE Part); BI 705564 10 mg fed/ BI 705564 10 mg fasted (FE Part)
Drug: BI 705564 (Reference) — Fasting state
  Arms: 1 milligram (mg) BI 705564 fasted (SRD part); 10 mg BI 705564 fasted (SRD part); 20 mg BI 705564 fasted (SRD part); 3 mg BI 705564 fasted (SRD part); 40 mg BI 705564 fasted (SRD part); 80 mg BI 705564 fasted (SRD part); BI 705564 10 mg fasted/ BI 705564 10 mg fed (FE Part); BI 705564 10 mg fed/ BI 705564 10 mg fasted (FE Part)

SUMMARY:
Investigation of safety, tolerability, pharmacokinetics and pharmacodynamics of single rising doses of BI 705564 and of the food effect on BI 705564 in healthy male subjects

DETAILED DESCRIPTION:
The primary objective of the single rising dose part under fasting and under fed conditions is to investigate safety and tolerability of BI 705564 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of pharmacokinetics (PK) including dose proportionality, and pharmacodynamics (PD) of BI 705564 after single rising doses.

The objective of the food effect part is to explore the relative bioavailability of BI 705564 tablets under fed and fasted conditions following the oral administration of single doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12 lead Electrocardiogram [ECG], and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body Mass Index [BMI] of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice [GCP] and local legislation

Exclusion Criteria:

-- Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator

* Repeated measurement of systolic blood pressure outside the range of 90 to 140mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/ or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication, if that might reasonably influence the results of the trial (incl. QT/ QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of the trial site
* A marked baseline prolongation of QT/ QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram [ECG] finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Male subjects with women of childbearing potential [WOCBP] partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Repeated absolute B cell (CD19+) counts below 40/μL at screening
* Repeated platelet counts below 100 cells/nL at screening
* Serum potassium below normal range at screening
* A history or current clinical signs of acute pancreatitis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a study in healthy men to test how different doses of BI 705564 are taken up in the body and whether taking BI 705564 with food makes a difference. The single rising dose (SRD) parts under fasting and fed conditions were designed as partially randomised within dose groups, placebo-controlled, single-blind, parallel-group design. The food effect (FE) part was designed as open-label, randomised, single-dose, two-period, two-sequence crossover design.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met. For the food effect part: Single dose for each treatment (2 single doses in total) were separated by a washout period of at least 10 days
Groups:
- Placebo Matching BI 705564 Fasted (SRD Part): Participants were administered single dose of placebo matching BI 705564 orally as powder for oral solution or film-coated tablet with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (h).
- Placebo Matching BI 705564 Fed (SRD Part): Participants were administered single dose of placebo matching BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- 1 Milligram (mg) BI 705564 Fasted (SRD Part): Participants were administered a single dose of 1 mg BI 705564 (4 milliliter x 0.25 milligram/milliliter (mg/mL)) orally from a reconstitution of powder for oral solution 20 mg with Solvent for Oral Solution 80 mL (HP-ß-Cyclodextrin 100 mg/mL) after an overnight fast of at least 10 h.
- 3 mg BI 705564 Fasted (SRD Part): Participants were administered a single dose of 3 mg BI 705564 (12 milliliter x 0.25 milligram/milliliter (mg/mL)) orally from a reconstitution of powder for oral solution 20 mg with Solvent for Oral Solution 80 mL (HP-ß-Cyclodextrin 100 mg/mL) after an overnight fast of at least 10 h.
- 10 mg BI 705564 Fasted (SRD Part): Participants were administered single dose of 1x10 mg (10 mg) BI 705564 orally as film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- 20 mg BI 705564 Fasted (SRD Part): Participants were administered single dose of 2x10 mg (20 mg) BI 705564 orally as film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- 40 mg BI 705564 Fasted (SRD Part): Participants were administered single dose of 4x10 mg (40 mg) BI 705564 orally as film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- 80 mg BI 705564 Fasted (SRD Part): Participants were administered single dose of 8x10 mg (80 mg) BI 705564 orally as film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- 20 mg BI 705564 Fed (SRD Part): Participants were administered single dose of 2x10 mg (20 mg) BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- 40 mg BI 705564 Fed (SRD Part): Participants were administered single dose of 4x10 mg (40 mg) BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- 80 mg BI 705564 Fed (SRD Part): Participants were administered single dose of 8x10 mg (80 mg) BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- 160 mg BI 705564 Fed (SRD Part): Participants were administered single dose of 1x100 mg and 6x10 mg (160 mg) BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- BI 705564 10 mg Fasted/ BI 705564 10 mg Fed (FE Part): Participants were administered single dose of 1x10 mg (10 mg) BI 705564 orally as film-coated tablet after an overnight fast of at least 10 h in period 1 (fast condition), with 240 milliliters (mL) of water.
  Followed by single dose of 1x10 mg (10 mg) BI 705564 after a high-fat, high-calorie meal in period 2 (fed condition). Both treatments were separated by a washout period of at least 10 days.
- BI 705564 10 mg Fed/BI 705564 10 mg Fasted (FE Part): Participants were administered single dose of 1x10 mg (10 mg) BI 705564 orally as film-coated tablet after a high-fat, high-calorie meal in period 1 (fed condition), with 240 milliliters (mL) of water.
  Followed by single dose of 1x10 mg (10 mg) BI 705564 after an overnight fast of at least 10 h in period 2 (fast condition). Both treatments were separated by a washout period of at least 10 days.
Period: Overall Study
Arm/Group | Placebo Matching BI 705564 Fasted (SRD Part) | Placebo Matching BI 705564 Fed (SRD Part) | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part) | BI 705564 10 mg Fasted/ BI 705564 10 mg Fed (FE Part) | BI 705564 10 mg Fed/BI 705564 10 mg Fasted (FE Part)
Started | 12 | 8 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 8 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 705564 Fasted (SRD Part) | Placebo Matching BI 705564 Fed (SRD Part) | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part) | BI 705564 10 mg Fasted/ BI 705564 10 mg Fed (FE Part) | BI 705564 10 mg Fed/BI 705564 10 mg Fasted (FE Part) | Total
Number analyzed (Participants) | 12 | 8 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (9.6) | 39.1 (6.1) | 36.0 (5.2) | 29.6 (8.4) | 32.5 (8.2) | 33.3 (9.3) | 36.8 (8.6) | 35.3 (8.6) | 37.7 (8.8) | 30.2 (6.7) | 33.8 (7.9) | 38.7 (7.6) | 29.3 (10.2) | 34.2 (12.2) | 34.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 8 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 8 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 91
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events (AEs)
Description: Number of participants with drug-related adverse events (AEs) is presented for SRD part.Percentage of participants with treatment-emergent drug-related Adverse Events (AEs) is reported.
  Percentages are calculated using total number of subjects per treatment as the denominator.
Time Frame: From drug administration until end of the treatment, up to 15 days (for SRD fasting and fed conditions).
Population: Treated set (TS): TS included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of the investigational treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Matching BI 705564 Total: Participants were administered single dose of placebo matching BI 705564 orally as powder for oral solution or film-coated tablet with 240 milliliters (mL) of water after an overnight fast of at least 10 h in fast condition or after a high-fat, high-calorie meal in fed condition.
- Total BI 705564 Fast (SRD Part): Participants were administered single dose of BI 705564 orally as powder for oral solution or film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- Total BI 705564 Fed (SRD Part): Participants were administered single dose of BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal
- Total BI 705564 (SRD Part): Participants were administered single dose of BI 705564 orally as powder for oral solution or film-coated tablet with 240 mL of water as after an overnight fast of at least 10 h in fast condition or after a high-fat, high-calorie meal in fed condition.
Arm/Group | Placebo Matching BI 705564 Fasted (SRD Part) | Placebo Matching BI 705564 Fed (SRD Part) | Placebo Matching BI 705564 Total | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | Total BI 705564 Fast (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part) | Total BI 705564 Fed (SRD Part) | Total BI 705564 (SRD Part)
Number analyzed (Participants) | 12 | 8 | 20 | 6 | 5 | 6 | 6 | 6 | 6 | 35 | 6 | 6 | 6 | 6 | 24 | 59
Participants | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 4 | 0 | 0 | 4 | 7

2. Primary Outcome: Area Under the Concentration-time Curve of BI 705564 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) (FE Part)
Description: AUC0-tz, area under the concentration-time curve of BI 705564 in plasma over the time interval from 0 to the last quantifiable data point for FE part is presented.
Time Frame: Pharmacokinetic samples were collected pre-dose and at 0:30 (hour: minute), 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 34:00, 48:00 and 72:00 after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): PKS included all subjects from the TS who provided at least 1 primary or secondary PK parameter (AUC0-∞ or Cmax) that was not excluded due to a protocol violation relevant to the evaluation of PK or due to non-evaluability.
Measure: Least Squares Mean (Standard Error); unit: nanomole*hour/litre [nmol*h/L]
Groups:
- 10 mg BI 705564 Fed (FE Part): Participants were administered single dose of 1x10 mg (10 mg) BI 705564 orally as film-coated tablet with 240 mL of water after a high-fat, high-calorie meal.
- 10 mg BI 705564 Fast (FE Part): Participants were administered single dose of 1x10 mg (10 mg) BI 705564 orally as film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
Arm/Group | 10 mg BI 705564 Fed (FE Part) | 10 mg BI 705564 Fast (FE Part)
Number analyzed (Participants) | 11 | 12
nanomole*hour/litre [nmol*h/L] | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 46.068. Standard error is actually geometric standard error. Geometric standard error ="1.099" | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 29.044. Standard error is actually geometric standard error. Geometric standard error =1.095
Statistical Analysis 1: Comparison: 10 mg BI 705564 Fed (FE Part) vs 10 mg BI 705564 Fast (FE Part); The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including effects for 'sequence', 'subjects nested within sequences', 'period' and 'treatment'. The effect "subjects within sequences" will be considered as random, the other effects as fixed; Test type: Other — No hypothesis was tested and no acceptance range was specified; Geometric mean (gMean) ratio (%) = 158.61, 90% CI 2-sided [133.679 to 188.195], Standard Error of Mean 22.4 — gMean ratio = 10 mg BI 705564 fed/10 mg BI 705564 fast. Standard Error of the mean is actually the intra-individual geometric coefficient variation

3. Primary Outcome: Maximum Measured Concentration of BI 705564 in Plasma (Cmax) (FE Part)
Description: Cmax, maximum measured concentration of BI 705564 in plasma is presented for FE part.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Nanomole/litre [nmol/L]
Arm/Group | 10 mg BI 705564 Fed (FE Part) | 10 mg BI 705564 Fast (FE Part)
Number analyzed (Participants) | 11 | 12
Nanomole/litre [nmol/L] | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 13.109 Standard error is actually geometric standard error. Geometric standard error =1.110 | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 6.751. Standard error is actually geometric standard error. Geometric standard error =1.105
Statistical Analysis 1: Comparison: 10 mg BI 705564 Fed (FE Part) vs 10 mg BI 705564 Fast (FE Part); [analysis description as in outcome 2, analysis 1]; Test type: Other — No hypothesis was tested and no acceptance range was specified; gMean ratio (%) = 194.18, 90% CI 2-sided [158.912 to 237.267], Standard Error of Mean 26.4 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Maximum Measured Concentration of BI 705564 in Plasma (Cmax) (SRD Part)
Description: Cmax, maximum measured concentration of BI 705564 in plasma is presented for SRD part.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole/litre [nmol/L]
Arm/Group | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Nanomole/litre [nmol/L] | 1.66 (26.9) | 7.51 (34.9) | 4.94 (25.9) | 12.9 (55.5) | 14.5 (40.7) | 16.5 (29.3) | 23.9 (17.0) | 41.2 (36.0) | 58.3 (12.1) | 122.0 (58.0)
Statistical Analysis 1: Comparison: 1 Milligram (mg) BI 705564 Fasted (SRD Part) vs 3 mg BI 705564 Fasted (SRD Part) vs 10 mg BI 705564 Fasted (SRD Part) vs 20 mg BI 705564 Fasted (SRD Part) vs 40 mg BI 705564 Fasted (SRD Part) vs 80 mg BI 705564 Fasted (SRD Part); The basic model for the investigation of dose proportionality for fasted condition was a power model that describes the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 0.4879, 95% CI 2-sided [0.3767 to 0.5990], Standard Error of Mean 0.0546 — Based on the estimate for slope parameter, a 2-sided 95% Confidence Interval (CI) for the slope was computed. Standard error of the mean is actually standard error of slope. Perfect dose proportionality would correspond to a slope of 1
Statistical Analysis 2: Comparison: 20 mg BI 705564 Fed (SRD Part) vs 40 mg BI 705564 Fed (SRD Part) vs 80 mg BI 705564 Fed (SRD Part) vs 160 mg BI 705564 Fed (SRD Part); The basic model for the investigation of dose proportionality for fed condition was a power model that describes the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 0.7553, 95% CI 2-sided [0.5736 to 0.9370], Standard Error of Mean 0.0876 — Based on the estimate for slope parameter, a 2-sided 95% CI for the slope was computed. Standard error of the mean is actually standard error of slope. Perfect dose proportionality would correspond to a slope of 1

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 705564 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (SRD Part)
Description: AUC0-∞, area under the concentration-time curve of BI 705564 in plasma over the time interval from 0 extrapolated to infinity is presented for SRD part.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/litre [nmol*h/L]
Arm/Group | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part)
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 5 | 6 | 6 | 4 | 5 | 6
nanomole*hour/litre [nmol*h/L] | NA (NA) — NA= Not calculated because plasma concentrations were below lower limit of quantification (BLQ) | NA (NA) — NA= Not calculated because plasma concentrations were below lower limit of quantification (BLQ) | NA (NA) — NA= Not calculated because plasma concentrations were below lower limit of quantification (BLQ) | 54.0 (29.7) | 74.2 (37.4) | 98.1 (43.4) | NA (NA) — NA= Not calculated because plasma concentrations were below lower limit of quantification (BLQ) | 185.0 (35.5) | 330.0 (31.2) | 481.0 (48.2)
Statistical Analysis 1: Comparison: 20 mg BI 705564 Fasted (SRD Part) vs 40 mg BI 705564 Fasted (SRD Part) vs 80 mg BI 705564 Fasted (SRD Part); [analysis description as in outcome 4, analysis 1]; Test type: Other; Slope = 0.4651, 95% CI 2-sided [0.1935 to 0.7368], Standard Error of Mean 0.1274 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: 40 mg BI 705564 Fed (SRD Part) vs 80 mg BI 705564 Fed (SRD Part) vs 160 mg BI 705564 Fed (SRD Part); [analysis description as in outcome 4, analysis 2]; Test type: Other; Power model; Slope = 0.6651, 95% CI 2-sided [0.3679 to 0.9622], Standard Error of Mean 0.1385 — [estimate comment as in outcome 4, analysis 2]

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 705564 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (FE Part)
Description: AUC0-∞, area under the concentration-time curve of BI 705564 in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 2
Population: PKS: Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/litre [nmol*h/L]
Arm/Group | 10 mg BI 705564 Fed (FE Part) | 10 mg BI 705564 Fast (FE Part)
Number analyzed (Participants) | 0 | 2
nanomole*hour/litre [nmol*h/L] |  | NA (NA) — Geometric mean and Geometric Coefficient of Variation could not be calculated because of the limited sample size.

ADVERSE EVENTS:
Time Frame: From drug administration until end of the treatment, up to 15 days (for SRD part fasting and fed condition and FE part).
Arm/Group | Placebo Matching BI 705564 Fasted (SRD Part) | Placebo Matching BI 705564 Fed (SRD Part) | Placebo Matching BI 705564 Total | 1 Milligram (mg) BI 705564 Fasted (SRD Part) | 3 mg BI 705564 Fasted (SRD Part) | 10 mg BI 705564 Fasted (SRD Part) | 20 mg BI 705564 Fasted (SRD Part) | 40 mg BI 705564 Fasted (SRD Part) | 80 mg BI 705564 Fasted (SRD Part) | Total BI 705564 Fast (SRD Part) | 20 mg BI 705564 Fed (SRD Part) | 40 mg BI 705564 Fed (SRD Part) | 80 mg BI 705564 Fed (SRD Part) | 160 mg BI 705564 Fed (SRD Part) | Total BI 705564 Fed (SRD Part) | Total BI 705564 (SRD Part) | 10 mg BI 705564 Fast (FE Part) | 10 mg BI 705564 Fed (FE Part)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/20 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/35 | 0/6 | 0/6 | 0/6 | 0/6 | 0/24 | 0/59 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/20 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/35 | 0/6 | 0/6 | 0/6 | 0/6 | 0/24 | 0/59 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 6/12 | 3/8 | 9/20 | 3/6 | 1/5 | 2/6 | 1/6 | 3/6 | 2/6 | 12/35 | 3/6 | 4/6 | 0/6 | 3/6 | 10/24 | 22/59 | 2/12 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 705564 Fasted (SRD Part) (N=12) | Placebo Matching BI 705564 Fed (SRD Part) (N=8) | Placebo Matching BI 705564 Total (N=20) | 1 Milligram (mg) BI 705564 Fasted (SRD Part) (N=6) | 3 mg BI 705564 Fasted (SRD Part) (N=5) | 10 mg BI 705564 Fasted (SRD Part) (N=6) | 20 mg BI 705564 Fasted (SRD Part) (N=6) | 40 mg BI 705564 Fasted (SRD Part) (N=6) | 80 mg BI 705564 Fasted (SRD Part) (N=6) | Total BI 705564 Fast (SRD Part) (N=35) | 20 mg BI 705564 Fed (SRD Part) (N=6) | 40 mg BI 705564 Fed (SRD Part) (N=6) | 80 mg BI 705564 Fed (SRD Part) (N=6) | 160 mg BI 705564 Fed (SRD Part) (N=6) | Total BI 705564 Fed (SRD Part) (N=24) | Total BI 705564 (SRD Part) (N=59) | 10 mg BI 705564 Fast (FE Part) (N=12) | 10 mg BI 705564 Fed (FE Part) (N=11)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 4 | 2 | 0 | 1 | 0 | 1 | 1 | 5 | 1 | 1 | 0 | 1 | 3 | 8 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT03123185/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03123185/SAP_001.pdf